CLINICAL TRIAL: NCT06233929
Title: Rheumatoid Arthritis Real-world Cohort Study in China (ReALSA)
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1235-01
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An ongoing long-term prospective cohort study is conducted by our team, that is dedicated to recruit patients with RA, to identify the development of clinical, biomedical, histopathological and imaging biomarkers for the diagnosis and prognosis of difficult-to-treat RA, and RA-related complications / comorbidities including sarcopenia, CVD, malignancies, specific infections (especially tuberculosis, herpes zoster, and HBV reactivation), and to evaluate their impact on the long-term prognosis of RA.

To improve the prognosis of RA, this study includes the following objectives:

1. Construct a useful database to explore the secular dynamic progress of RA, including RA progression and complications (e.g., sarcopenia, CVD, malignancies, infections), as well as to improve our understanding of the life-course factors affecting the process that will facilitate future research activities.
2. Identify the potential biomarkers (clinical, biochemical, histopathological, and imaging markers) to develop multimodal models predicting outcomes in high-risk RA subgroups like difficult-to-treat RA.
3. Develop the related multi-modal prediction models with clinical, biomedical and imaging variables to improve the diagnosis and prognosis of RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older and diagnosed with RA according to 1987 ACR or 2010 ACR / EULAR classification criteria

Exclusion Criteria:

* Patients do not plan to receive long-term healthcare at SYSMH, PYCH or SS-SYSMH
* Patients unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with RA will be consecutively recruited during 2024 and 2033 from the Department of Rheumatology, Sun Yat-sen Memorial Hospital (SYSMH) of Sun Yat-sen University, The Affiliated Panyu Central Hospital (PYCH) of Guangzhou Medical University in Guangzhou, and ShenShan Medical center, Memorial Hospital of Sun Yat-sen University (SS-SYSMH) in Shanwei, P.R China. The inclusion criteria for this study are as follows: 1) diagnosis with RA according to 1987 ACR [41] or 2010 ACR/EULAR classification criteria [42]; 2) age ≥ 18 years old. The exclusion criteria are as follows: 1) patients do not plan to receive long-term healthcare at SYSMH, PYCH or SS-SYSMH; 2) unable to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
RA disease outcomes | 60 months
  The primary clinical end-point is the proportion of patients achieving CDAI remission (CDAI≤2.8). The primary functional end-point is the proportion of patients with functional limitation (HAQ-DI>1) . The primary radiographic end-point is the proportion of patients without radiographic progression defined as no increase in mTSS from baseline to 60 months (ΔmTSS≤0) . Radiographs are scored by two experienced and well-trained readers (a radiologist and a rheumatologist) who are aware of the chronological order of the sets of images but not unaware of all other data .
RA-related complication or comorbidity outcomes | All adverse events are collected from the time the subject signs the informed consent form until the end of the follow-up period
  Predefined RA-related complication or comorbidity end-points are muscular, cardiovascular, malignant, specific infectious outcomes and additional adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology, Sun Yat-sen Memorial Hospital (SYSMH) of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin JZ, Zhu Y, Li QH, Ouyang ZM, Liu HJ, Zou YW, Yang Y, Yang KM, Yang LJ, Yang ZH, Zhang L, Mo YQ, Ma JD, Dai L. Rheumatoid Arthritis Real-world Cohort Study in China (ReALSA): protocol for a multicentre prospective, longitudinal cohort study. BMJ Open. 2025 Jul 13;15(7):e092583. doi: 10.1136/bmjopen-2024-092583. PMID 40659397